CLINICAL TRIAL: NCT00634218
Title: REaching and Treating LGBT Smokers: The Internet
Brief Title: Reaching and Treating Lesbian, Gay, Bisexual, and Transgender (LGBT) Cigarette Smokers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Principal Investigator, Gary Humfleet, Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TRDRP 15RT-0165
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Cigarette Smoking
Keywords: nicotine; smoking; smoking cessation
MeSH Terms: conditions — Cigarette Smoking; Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Mail-based Self Help (MSH) treatment. Participants will receive the self-help manual developed specifically for LGBT smokers.
  Interventions: Behavioral: Self-Help Manual
- 2 (Active Comparator): Mail-based Self Help plus an Internet-based Smoking Treatment (IST). In the IST condition, participants will receive the manual plus access to an Internet-based intervention that includes social support.
  Interventions: Behavioral: Mail-based Self-help plus Internet-based Smoking Treatment
- 3 (Active Comparator): Mail-based Self-Help plus Telephone Counseling (TC). In the TC condition, participants will receive a self-help manual specifically developed for LGBT smokers plus 6 telephone-based counseling sessions.
  Interventions: Behavioral: Self-Help Manual plus Telephone counseling
- 4 (Active Comparator): Mail-based Self-Help plus an Internet-based Intervention plus Telephone Counseling. Participants will receive a self-help manual, have access to an internet-based smoking treatment and participante in 6 telephone counseling sessions.
  Interventions: Behavioral: Self-Help Manual plus Internet-based Intervention plus Telephone Counseling

INTERVENTIONS:
Behavioral: Mail-based Self-help plus Internet-based Smoking Treatment — Participants in this condition will received a self-help manual developed specifically for LGBT smokers and access to an Internet-based smoking cessation treatment program. The website provides education and information about smoking cessation alond with development of a personalized quit plan. Participants have access to a message board where they can contact other participants.
  Arms: 2
Behavioral: Self-Help Manual plus Telephone counseling — Participants will receive a self-help manual specifically developed for LGBT smokers plus 6 telephone-based counseling sessions. The counseling sessions focus on the development of a personalized plan to quit smoking and occur over a 3 month period.
  Arms: 3
Behavioral: Self-Help Manual — Participants will receive a self-help smoking cessation manual specifically developed for LGBT smokers. The manual provides information on quitting smoking and encourages the development of a personalized quit plan through various activities and exercises.
  Arms: 1
Behavioral: Self-Help Manual plus Internet-based Intervention plus Telephone Counseling — Participants in this condition will received a self-help manual developed specifically for LGBT smokers and access to an Internet-based smoking cessation treatment program. The website provides education and information about smoking cessation alond with development of a personalized quit plan. Participants have access to a message board where they can contact other participants. Smokers will also receive 6 telephone-based counseling sessions which occur over a 3 month period
  Arms: 4

SUMMARY:
Smoking rates are significantly higher among lesbian, gay, bisexual, and transgender (LGBT) populations compared to the general population. LGBT individuals may be at increased risk for experiencing psychosocial issues, e.g., negative moods, stress, alcohol/drug use, that have been associated with smoking treatment failure in other groups of smokers. Technology, such as the Internet and telephone, can be an effective method to reach a large number of smokers and may be particularly effective in reaching hidden populations. Thus, the study seeks to examine whether Internet-based counseling and/or telephone counseling can improve quit rates for LGBT smokers.

Participants (N=600) will be randomly assigned to one of four conditions: 1) a Mail-based Self Help (MSH) treatment; 2) MSH plus an Internet-based Smoking Treatment (IST); MSH plus Telephone Counseling (TC) or 4) MSH plus IST plus TC. Participants in the MSH condition will receive a self-help smoking cessation manual. In the IST condition, participants will receive the manual plus access to an Internet-based intervention that includes social support. In the TC condition, participants will receive the manual plus 6 telephone-based counseling sessions. In the fourth condition, participants will receive the manual plus access to an Internet-based intervention plus telephone counseling. Before starting treatment, participants will complete questionnaires on smoking, nicotine dependence, demographics, negative mood, and alcohol use. Participants will be contacted at 3, 6, and 12 months after enrollment to determine whether they are smoking. The data will be analyzed to compare the efficacy of the four treatments and to examine the possible influence of existing social networks and level of negative mood on treatment outcome and to examine the possible influence of residency (rural versus urban) on use of the Internet-based treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* identify as lesbian, gay, bisexual, or transgender
* access to the internet
* valid email account
* valid telephone number
* English speaking
* resident of the U.S.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Smoking status | 3,6, and 12 months following enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of California, San Francisco, San Francisco, California, United States